CLINICAL TRIAL: NCT04455594
Title: Almonertinib Vs. Erlotinib/Chemotherapy for Neo-adjuVant Treatment of Stage IIIA-N2 EGFR-mutated NSCLC: a Multicenter, Open-label, Phase II Randomized Controlled Trial
Brief Title: Almonertinib Vs. Erlotinib/Chemotherapy for Neo-adjuVant Treatment of Stage IIIA-N2 EGFR-mutated NSCLC
Acronym: ANSWER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Chief Surgeon, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-LK-2020-005
Record Dates: First submitted 2020-06-19; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Non-Small Cell Lung Cancer Stage IIIA
Keywords: resectable NSCLC, IIIA-N2 NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Erlotinib Hydrochloride; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib (Experimental): Almonertinib 110mg QD
  Interventions: Drug: Almonertinib
- Investigator-choice therapy (Erlotinib or Chemotherapy) (Active Comparator): Erlotinib 150mg QD or Cisplatin(75mg/m2) or Carboplatin (AUC=5) to be administered with pemetrexed (500mg/m2) on Day 1 of every 3-week cycle for 3 cycles
  Interventions: Drug: Erlotinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Almonertinib — Oral, 110mg QD
  Other Names: HS-10296
  Arms: Almonertinib
Drug: Erlotinib — Oral, 150mg QD
  Arms: Investigator-choice therapy (Erlotinib or Chemotherapy)
Drug: Cisplatin — Cisplatin(75mg/m2) be administered with pemetrexed (500mg/m2) on Day 1 of every 3-week cycle for 3 cycles
  Arms: Investigator-choice therapy (Erlotinib or Chemotherapy)
Drug: Carboplatin — Carboplatin (AUC=5) to be administered with pemetrexed (500mg/m2) on Day 1 of every 3-week cycle for 3 cycles
  Arms: Investigator-choice therapy (Erlotinib or Chemotherapy)
Drug: Pemetrexed — Pemetrexed (500mg/m2) to be administered with Cisplatin(75mg/m2) or Carboplatin (AUC=5) on Day 1 of every 3-week cycle for 3 cycles
  Arms: Investigator-choice therapy (Erlotinib or Chemotherapy)

SUMMARY:
This is a multicenter, randomized, controlled, phase II study assessing the efficacy and safety of Almonertinib compared Erlotinib or platinum doublet chemotherapy (carboplatin or cisplatin + pemetrexed) as neoadjuvant therapy to EGFRm+ IIIA-N2 NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age at least 18 years, no more than 75 years.
2. Previously untreated, histologically documented NSCLC with completely or potentially resectable IIIA-N2 nonsquamous NSCLC(according to Version 8 of AJCC staging). N2 is defined as as radiologically and pathologically confirmed, nonbulky metastases to single-station mediastinal lymph nodes (lymph nodes < 2 cm in short axis) that are expected to be completely resectable.
3. Tumor tissue samples or blood samples are confirmed as EGFR sensitive mutations by central laboratory tests (including Ex19del or L858R, both alone or with other EGFR mutations). If the tumor tissue is accessible, the tumor tissue is recommended to be submitted for examination. If tumor tissue is not accessible or patient cannot undergo tissue biopsy, blood sample is also allowed.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
5. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as >= 10 mm in the longest diameter (except lymph nodes, which must have short axis >= 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and baseline tumour assessment scans are done at least 14days afar the screening biopsy is performed.
6. Women of childbearing potential must use a contraception method during the study treatment and for at least 3 months after the treatment is completed; must have a negative pregnancy test prior to starting treatment or proved no risk of pregancy by meeting one of the following criteria:

   1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
   3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
7. Male patients should be willing to use barrier contraception (i.e., condoms) during the study treatment and for at least 3 months after the treatment is completed.
8. Signed and dated informed consent form.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Prior surgical resection of lung cancer.
   2. Prior treatment with any EGFR TKI.
   3. Prior treatment with any chemotherapy for NSCLC
   4. Prior treatment with any radiotherapy for NSCLC
   5. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   6. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.
2. Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of study drug.
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy.
4. Patients with malignant pleural effusion. [only exception: pleural effusion on CT scan (not visible on CXR) or considered too small and pericardial effusion]
5. Patients who received yellow-fever vaccine or other attenuated live vaccine during pemetrexed treatment.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required.
7. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Almonertinib.
8. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) <= 40%.
9. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
10. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count (ANC) < 1.5 x 10^9 / L;
    2. Platelet count <100 x 10^9 / L;
    3. Hemoglobin < 90 g/L (<9 g/dL);
    4. Alanine aminotransferase > 2.5 x upper limit of normal (ULN).
    5. Aspartate aminotransferase (AST) > 2.5 x ULN.
    6. Total bilirubin (TBL) > 1.5 x ULN or > 3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia).
    7. Creatinine > 1.5 x ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 x ULN.
11. Women at breastfeeding or have a negative serum or urine pregnancy test in the 3 days prior to the start of the treatment..
12. History of hypersensitivity to any active or inactive ingredient of Almonertinib, or to drugs with a similar chemical structure or class to Almonertinib.
13. History of hypersensitivity to any active or inactive ingredient of Erlotinib, or to drugs with a similar chemical structure or class to Erlotinib.
14. With lactose in the tablets, patients with rare genetic disease like galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not use use erlotinib.
15. Patients who are allergic to pemetrexed or any other component of the preparation, carboplatin or cisplatin.
16. Patients with contraindications of pemetrexed and carboplatin or cisplatin.
17. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
18. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
19. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of randomization to an average of 6 weeks after the first dose
  Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.

SECONDARY OUTCOMES:
Pathological complete response (pCR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as absence of any residual cancer cells in the surgical specimen assessed post-surgery
Major Pathological Response (MPR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as ≤10% residual cancer cells in the surgical specimen, as assessed per central pathology laboratory post-surgery
Disease free survival (DFS) | From date of randomization up to approximately 18 months after date of resection
  DFS is defined as the time from the date of surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.
  If there is residual disease after surgery (eg. positive margins), the DFS event is the date of surgery.
Overall Survival (OS) | Up to approximately 5.5 years after the last patient is randomized
  Patients will be followed up to approximately 5.5 years after they are randomized.
R0 resection rate | Up to 1 week after surgery
Downstaging rate | From date of randomization to an average of 12 weeks after the first dose
  Measured using lymph node staging
Concordance of EGFRm status between plasma-derived ctDNA | Baseline, up to 1 week before surgery and up to 1 week after surgery
Incidence of Adverse Events (AEs) | Up to 80 weeks
  According to CTCAE4.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China